CLINICAL TRIAL: NCT06444334
Title: Evaluation of the Effect of Laser Biostimulation on Implant Covered With PRF in Controlled Diabetic Patients: A Randomized Clinical Trial
Brief Title: Laser Biostimulation on Implant Covered With PRF in Controlled Diabetics
Acronym: PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Said Abd Allah Kamel Taha, Principal investigator, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 03430423
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Diabetes; Implant Site Reaction; Platelet Rich Fibrin
Keywords: laser biostimulation; PRF; implants; osseointegration; diabetic patient
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: 22 implants were divided randomly into 2 groups. Group1: control group (no laser irradiation), group2: diode laser irradiation group
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the participants as in group 1 or control laser device is off (not active)while in group 2 laser device is active. Outcome Assessor is blinded as the cases is coded and unknown for the Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control PRF group (Active Comparator): controlled diabetic patients with 11 implants covered with PRF inserted in posterior maxilla or mandible, not laser irradiated
  Interventions: Procedure: PRF platelet rich fibrin
- laser and PRF test group (Experimental): controlled diabetic patients with 11 implants covered with PRF inserted in posterior maxilla or mandible, expoed to Diode laser irradiation
  Interventions: Radiation: low level Diode Laser; Procedure: PRF platelet rich fibrin

INTERVENTIONS:
Radiation: low level Diode Laser — Group 2 was exposed to laser irradiation following implant insertion for 3 sessions: Immediately after implant insertion, 2 days after implant insertion and 1 week after insertion , using a red Diode(gallium-aluminun-arsenide) LLLT using calibrated diode laser device
  Arms: laser and PRF test group
Procedure: PRF platelet rich fibrin — The preparation method of PRF was performed in accordance with the protocol developed by Choukroun et al 2001. PRF was withdrawn and processed from the same operated-on patient's blood; 6ml IV blood withdrawn from the antecubital vein in to two sterile 3ml red vacutainer tubes without anticoagulant, followed by a 12 minute centrifuge with 3000 RPM producing a platelet rich fibrin clot, which is then incised & separated with 2mm basal layer of RBCs rich in growth factors

SUMMARY:
the goal of this clinical trial is to evaluate laser biostimulation effect on osseointegration of implant covered by PRF(platelet rich fibrin) in controlled diabetic patients with compromised healing potential.

METHODS: The study was conducted on type 2 controlled diabetic patients receiving 22 implants covered with PRF inserted in posterior maxilla or mandible. Implants were divided randomly into 2 groups. Group1: control group (received no laser irradiation), group2: received diode laser. Peri-implant new bone density and secondary stability were assessed using cone-beam computed tomography and Anycheck device respectively. Density was evaluated immediately post implant insertion and after 5 months, while implant stability was performed 5 months post implant insertion. Statistical analysis was executed significance level P ≤ 0.05.

DETAILED DESCRIPTION:
Study type:

randomized controlled clinical trial.

Study design:

Controlled type II diabetic patients with edentulous posterior areas were randomly selected from dental clinic of Medical and Scientific Centre of Excellence (MSCE), National Research Centre (NRC), Cairo, Egypt, according to inclusion and exclusion criteria to receive a total number of twenty-two dental implants. Implants were randomly distributed with 1:1 allocation ratio into two groups according to exposure to laser irradiation. Group 1 was not exposed to laser irradiation (control group), while group 2 was exposed to laser irradiation. Peri-implant new bone density was evaluated immediately post implant insertion and after 5 months, while secondary implant stability was performed 5 months post implant insertion.

This study was prosecuted with the Code of Ethics of the World Medical Association, they were stated in the Declaration of Helsinki in 1975. Medical Research Ethical Committee of the National Research Centre, Cairo, Egypt permitted this study with approval number (03430423). All patients were familiar with the study's treatment phases and signed a consent form. The study was conducted from January 2023 to March 2024

Radiographic procedures:

Every patient had undergone radiographic analysis pre-operatively using cone beam computed tomography (CBCT) . The intended size and location of the implants were determined and planned virtually by digital software (Planmeca Romexis Viewer 6.2.1.19). Bone density around the implants will be evaluated using CBCT software at (immediately postoperative as baseline and 5 months postoperative. Both groups were radiographed by cone beam CT for evaluation and assessment of bone density around implants by professional blinded investigators. Planmeca Romaxies machine was used with the following specifications: Field of View (FOV) = 8.0x5.0 cm, resolution = 0.300, orientation = portrait, 90 kV, 80mA, and exposure time = 15.019 sec.

Surgical procedures:

Implants (K1 line conical connection double thread, OXY, Italy) were inserted under profound local anesthesia using free hand open flap technique; where mucoperiosteal gingival envelop full thickness flap was performed by crestal incision & mucoperiosteal reflection exposing bone . The preplanned location was confirmed by the aid of CBCT, then sequential drilling was exerted using graduated drills with stoppers under copious amount of saline coolant with the aid of paralleling pins if multiple implants were inserted to be splinted in the same patient.

Implants were screwed with torque between 35-45N to ensure primary stability. Various implants' sizes were utilized ranging from 4 mm to 5.5mm in diameter and from 8mm to 11mm in length in accordance with the virtual pre-plan based on bone geometrical availability. The procedure was executed by a single well-experienced operator who was blinded to the groups.

PRF preparation protocol:

The preparation method of PRF was performed in accordance with the protocol developed by Choukroun. PRF was withdrawn and processed from the same operated-on patient's blood; 6ml IV blood withdrawn from the antecubital vein in to two sterile 3ml red vacutainer tubes without anticoagulant, followed by a 12 minute centrifuge with 3000 RPM producing a platelet rich fibrin clot, which is then incised & separated with 2mm basal layer of RBCs rich in growth factors . Following the cover screw placement, PRF was extended bucco-lingually and mesio-distally over the alveolar ridge . Finally, approximation of the flap was achieved using non-resorbable 3/0 suture which was removed after 7-10 days postoperative. Nonsteroidal anti-inflammatory drugs and antibiotics were administered for seven days. Delayed loading was initiated after 5 months of osseointegration process.

Laser irradiation protocol:

Group 2 was exposed to laser irradiation following implant insertion for 3 sessions: Immediately after implant insertion, 2 days after implant insertion and 1 week after insertion , using a red Diode(gallium-aluminum-arsenide) LLLT using calibrated diode laser device at 635nm wavelength delivered by biomodulating handpiece with the following set parameters: 100mw power output, 8mm handpiece diameter, continuous mode, and time 40 second per point and contact mode . The laser probe was directed towards the implant site, gently touching the tissues mesially, distally, buccally, and lingually to assure the full exposure of the target surface to laser beam.

ELIGIBILITY:
Inclusion Criteria:

1. nonsmoker patients,
2. age range 30 -60 years,
3. Glycosylated hemoglobin (Hb1C) ranges between 7-8,
4. no other systemic disease,
5. vital signs are normal (blood pressure, temperature, pulse rate, respiratory rate),
6. missing 1st or 2nd mandibular or maxillary premolars or molars,
7. lab investigations are within normal (CBC. liver function AST &ALT, kidney function urea &creatinine, Ca level, 25OH Vit D),
8. no need for alveolar bone grafting, and
9. no soft or hard tissue pathology.

Exclusion Criteria:

1. smoker patient,
2. Glycosylated hemoglobin (Hb1C) more than 8 or less than 7,
3. age less than 30 or more than 60,
4. presence of other systemic diseases,
5. vital signs are not normal,
6. lab investigations are not normal (CBC, liver function, kidney function),
7. need for alveolar bone grafting and
8. present soft or hard tissue pathology.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Per-implant bone density measurements | at immediate day of surgery(baseline) and after 5 months for the same patients
  Digital software program was used for quantitative mean bone density measurements of all the captured radiographs produced by CBCT for both groups. Multiplanar resolution screen (MPR) was selected showing radiographic images of the mandible and maxilla in sagittal and coronal views to quantify bone radiodensity in mesiodistal and buccolingual surfaces respectively , a constant exact area was selected for each view with area =1 5.2mm2, width = 2.00mm, and height = 7.60mm. Five readings of radiodensity in Hounsfield units (HU statistics) were collected by blind investigator for each peri-implant surface (mesial, distal, buccal, and lingual) with slice thickness of 0.5mm. Finally, the mean density values were calculated and tabulated concerning sagittal and coronal views in each implant

SECONDARY OUTCOMES:
Implant stability measurements | only after 5 months from implant insertion
  AnyCheck device (AnyCheck, Neobiotech Co., Ltd. E-space #1001, 36, Digital-ro 27-gil, Guro-gu, Seoul, Korea, 08381) was utilized 5 months (2nd stability) post implant insertion. AnyCheck is an implant stability meter that measures the stiffness of the alveolar bone-implant interface through a tapping-motion. The degree of osseointegration is calculated in terms of IST (Initial Stability Test) value between 30 to 85. AnyCheck was turned on, then, the tip of the tap¬ping rod maintained contact angle between 0 to 30 degrees with healing abutment. The START button was gently pressed while holding the device stable, the measured value displayed on the LCD screen was recorded. The smaller the measured value, the weaker the degree of osseointegration. Mesiodistal and buccolingual sides of the implant were measured, five IST readings for each side were repetitively recorded by blind examiner and the mean reading was calculated and tabulated

CONTACTS AND LOCATIONS:
Overall Officials: Noha M Ismael, PhD, Study Director — National Research Centre, Egypt
Locations (1):
- Oral Surgery Clinic at National Research Centre, Giza, Egypt

REFERENCES:
- [Background] ELsyad MA, Abdraboh AE, Aboelnagga MM, Ghali RM, Lebshtien IT. Effect of Low-Level Laser Irradiation on Stability and Marginal Bone of Narrow Implants Retaining Overdentures in Moderately Controlled Diabetic Patients. J Oral Implantol. 2019 Oct;45(5):391-397. doi: 10.1563/aaid-joi-D-18-00263. Epub 2019 Aug 7. PMID 31389750
- [Background] Naujokat H, Kunzendorf B, Wiltfang J. Dental implants and diabetes mellitus-a systematic review. Int J Implant Dent. 2016 Dec;2(1):5. doi: 10.1186/s40729-016-0038-2. Epub 2016 Feb 11. PMID 27747697
- [Background] Taha SK, El Fattah SA, Said E, Abdel-Hamid MA, Nemat AH, El Shenawy H. Effect of Laser Bio-Stimulation on Mandibular Distraction Osteogenesis: An Experimental Study. J Oral Maxillofac Surg. 2018 Nov;76(11):2411-2421. doi: 10.1016/j.joms.2018.04.030. Epub 2018 May 7. PMID 29856939
- [Background] 4. El-banna R, Shafik M, Shoreibah E: Effect of Platelet Rich Fibrin on the Healing of Intra-bony Defects: A Clinical Study. ADJ-for Girls, Vol. 5, No. 1, January (2018) - PP. 29:35 doi10.21608/adjg.2018.7990
- [Background] 5.Ghazal, Asmaa M.; Hassan, Susan H.; Mohamed, Fatma I.; Namat, Amany H.; and Taha, Said K. (2023)
- [Background] 6.Allam AF, Zaky AA, Elshenawy HM, Safwat EM, Hassan ML, Nassar MA, Taha, S.K: Evaluating The Biostimulation Effect Of Diode Laser 650 Nm Combined With TEMPO Oxidized Nano-Cellulose Mixed With Biphasic Tricalcium Phosphate On Bone Healing: Experimental Animal Study. Journal of pharmaceutical Negative Results ¦ Volume 14 ¦ Special Issue 2 ¦ 2023
- [Background] Khorshidi H, Raoofi S, Bagheri R, Banihashemi H. Comparison of the Mechanical Properties of Early Leukocyte- and Platelet-Rich Fibrin versus PRGF/Endoret Membranes. Int J Dent. 2016;2016:1849207. doi: 10.1155/2016/1849207. Epub 2016 Jan 6. PMID 26880919
- [Background] 8-Mowla AE, Sherif H, Bashir D. Evaluation of the effect of platelet rich fibrin (PRF) on bone regeneration in the tibia of diabetic rats (histological and immunohistochemical studies). Egypt J Histol.2020; 43(3): 777-790.
- [Background] Mayer L, Gomes FV, de Oliveira MG, de Moraes JF, Carlsson L. Peri-implant osseointegration after low-level laser therapy: micro-computed tomography and resonance frequency analysis in an animal model. Lasers Med Sci. 2016 Dec;31(9):1789-1795. doi: 10.1007/s10103-016-2051-3. Epub 2016 Aug 17. PMID 27534769
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] 11- Choukroun J AF,Schoeffler C, Vervelle A. Une opportunite en paro-implantologie:Le PRF.Implantodontie2001;42:55-62
- [Background] Matys J, Swider K, Grzech-Lesniak K, Dominiak M, Romeo U. Photobiomodulation by a 635nm Diode Laser on Peri-Implant Bone: Primary and Secondary Stability and Bone Density Analysis-A Randomized Clinical Trial. Biomed Res Int. 2019 Apr 22;2019:2785302. doi: 10.1155/2019/2785302. eCollection 2019. PMID 31143771
- [Background] Dos Santos RG, Santos GS, Alkass N, Chiesa TL, Azzini GO, da Fonseca LF, Dos Santos AF, Rodrigues BL, Mosaner T, Lana JF. The regenerative mechanisms of platelet-rich plasma: A review. Cytokine. 2021 Aug;144:155560. doi: 10.1016/j.cyto.2021.155560. Epub 2021 May 15. PMID 34004552
- [Background] Habash G, Jayash SN. Diode laser assisted horizontal bone defect regeneration in the treatment of peri-implantitis. Clin Case Rep. 2021 Jan 3;9(3):1247-1252. doi: 10.1002/ccr3.3741. eCollection 2021 Mar. PMID 33768820
- [Background] 15- El-banna R, Shafik M, Shoreibah E, Zouair M,Adel Hamid M: Effect of Platelet Rich Fibrin on the Healing of Intra-bony Defects: A Clinical and Experimental Study. Dissertation, faculty of dental Medicine -Al Azhar University 2017
- [Background] Karaca IR, Ergun G, Ozturk DN. Is Low-level laser therapy and gaseous ozone application effective on osseointegration of immediately loaded implants? Niger J Clin Pract. 2018 Jun;21(6):703-710. doi: 10.4103/njcp.njcp_82_17. PMID 29888715
- [Background] Arakeeb MAA, Zaky AA, Harhash TA, Salem WS, El-Mofty M. Effect of Combined Application of Growth Factors and Diode Laser Bio-Stimulation on the Osseo Integration of Dental Implants. Open Access Maced J Med Sci. 2019 Aug 12;7(15):2520-2527. doi: 10.3889/oamjms.2019.672. eCollection 2019 Aug 15. PMID 31666858
- [Background] Sleem SSMEB, Zayet MK, El-Ghareeb TI, Saleh HAK. Evaluation of The Bio-Stimulatory Effect of Platelet Rich Fibrin Augmented by Diode LASER Compared to Platelet Rich Fibrin Alone on Dental Implant Replacing Posterior Mandibular Teeth. Randomised Clinical Trial: Split Mouth Study. Open Access Maced J Med Sci. 2019 Mar 14;7(5):869-875. doi: 10.3889/oamjms.2019.183. eCollection 2019 Mar 15. PMID 30962853
- [Background] Soares LG, Magalhaes EB, Magalhaes CA, Ferreira CF, Marques AM, Pinheiro AL. New bone formation around implants inserted on autologous and xenografts irradiated or not with IR laser light: a histomorphometric study in rabbits. Braz Dent J. 2013;24(3):218-23. doi: 10.1590/0103-6440201302186. PMID 23969909
- [Background] Batista JD, Sargenti-Neto S, Dechichi P, Rocha FS, Pagnoncelli RM. Low-level laser therapy on bone repair: is there any effect outside the irradiated field? Lasers Med Sci. 2015 Jul;30(5):1569-74. doi: 10.1007/s10103-015-1752-3. Epub 2015 May 15. PMID 25975746
- [Background] Mandic B, Lazic Z, Markovic A, Mandic B, Mandic M, Djinic A, Milicic B. Influence of postoperative low-level laser therapy on the osseointegration of self-tapping implants in the posterior maxilla: a 6-week split-mouth clinical study. Vojnosanit Pregl. 2015 Mar;72(3):233-40. doi: 10.2298/vsp131202075m. PMID 25958474
- [Background] Kusek ER. Immediate implant placement into infected sites: bacterial studies of the Hydroacoustic effects of the YSGG laser. J Oral Implantol. 2011 Mar;37 Spec No:205-11. doi: 10.1563/AAID-JOI-D-10-00014. Epub 2010 Aug 16. PMID 20712437
- [Background] Buser D, Weber HP, Lang NP. Tissue integration of non-submerged implants. 1-year results of a prospective study with 100 ITI hollow-cylinder and hollow-screw implants. Clin Oral Implants Res. 1990 Dec;1(1):33-40. doi: 10.1034/j.1600-0501.1990.010105.x. PMID 2099210